CLINICAL TRIAL: NCT05938764
Title: An Open-Label, Pilot-Feasibility Randomized Controlled Trial of Motivational Interviewing and the Community Reinforcement Approach With a Southwest Tribe
Brief Title: A Randomized Controlled Trial of Culturally Adapted Evidence-based Treatment With a Southwest Tribe
Acronym: MICRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-235; R01DA021672 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2023-07-10 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Substance Use Disorders
Keywords: Addiction treatment outcome; American Indian/Alaska Native; Indigenous; randomized controlled trial; Motivational Interviewing; Community Reinforcement Approach; Substance Use Disorder; Cultural Adaptation
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two phases: Phase one: a feasibility (N = 9) non-randomized, one-group design wherein all participants received culturally adapted Motivational Interviewing and Community Reinforcement Approach (MICRA) Phase two: This study used a mixed efficacy/effectiveness (hybrid) randomized controlled trial of two treatment arms (Treatment as usual-TAU and Motivational Interviewing and Community Reinforcement Approach-MICRA) with a parallel design and follow-up assessments at 4-, 8-, and 12-months post baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing and Community Reinforcement Approach (Active Comparator): A psychosocial intervention culturally tailoring the combination of motivational interviewing (approximately 1-3 individual therapy sessions) and the community reinforcement approach (could include maximum range of 15-19 individual therapy sessions). Two tribal members were hired and trained to deliver this intervention and were located separately from the other arm.
  Interventions: Behavioral: MICRA
- Treatment as Usual (Active Comparator): Treatment as usual (TAU) included an intake session and could include individual counseling, group counseling, or cultural education. Treatment as usual was provided by staff at the reservation based outpatient treatment center. There was no limit on number of sessions provided.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: MICRA — see earlier description
  Other Names: culturally adapted motivational interviewing and community reinforcement approach
  Arms: Motivational Interviewing and Community Reinforcement Approach
Behavioral: TAU — see earlier description
  Other Names: Treatment As Usual
  Arms: Treatment as Usual

SUMMARY:
This study combined, adapted and tested motivational interviewing (MI) and the Community Reinforcement Approach (CRA) as a culturally congruent treatment approach for Native Americans. This pilot-feasibility research was conducted in collaboration with a Southwest Tribe. The specific aims of this project were: Aim 1. To develop, in collaboration with the Tribal community, a combination of MI and CRA (MICRA) that is culturally adapted and includes a secondary focus on HIV/STD prevention; Aim 2. To develop and field test culturally-congruent research materials and procedures; Aim 3. To train Tribal behavioral health professionals in delivery of MICRA, and test (N=9) procedures for MICRA certification, supervision, and fidelity assurance; Aim 4. To conduct a pilot study (N=79) to estimate effect sizes for MICRA on key outcome variables with participants; and Aim 5. To estimate the types and prevalence of emotional distress and psychological and health problems likely to be encountered when treating substance use disorders in Native American populations.

MICRA Project was conducted in two phases: Phase 1 was a feasibility (N = 9) non-randomized one-group design wherein all participants received culturally adapted MICRA.

Phase 2 was a pilot (N = 79) comparing the effectiveness of MICRA and TAU. Following the screening and baseline interview, participants were randomized to receive MICRA or treatment as usual (TAU). Participants randomized to MICRA could receive up to a maximum of 16 to 20 therapy sessions with one of the MICRA counselors over the course of 16 weeks. In TAU, participants received standard outpatient services at the Tribal substance use disorder treatment center.

The primary hypotheses were: (1) the feasibility test (N=9) would yield improved percent days abstinent from all substances (excluding tobacco) from baseline to the 8-month follow-up, and (2) In the pilot randomized controlled trial of MICRA versus treatment as usual (TAU), the investigators hypothesized that percent days abstinent from all substances would be greater at the 12-month follow-up timepoint compared to TAU.

DETAILED DESCRIPTION:
This study combined, adapted and tested motivational interviewing (MI) and the Community Reinforcement Approach (CRA) as a culturally congruent treatment approach for Native Americans. This pilot-feasibility research was conducted in collaboration with a Southwest Tribe. The specific aims of this project were: Aim 1. To develop, in collaboration with the Tribal community, a combination of MI and CRA (MICRA) that is culturally adapted and includes a secondary focus on Human Immunodeficiency Virus / sexually transmitted disease (HIV/STD) prevention; Aim 2. To develop and field test culturally-congruent research materials and procedures; Aim 3. To train Tribal behavioral health professionals in delivery of MICRA, and test (N=9) procedures for MICRA certification, supervision, and fidelity assurance; Aim 4. To conduct a pilot study (N=79) to estimate effect sizes for MICRA on key outcome variables with participants; and Aim 5. To estimate the types and prevalence of emotional distress and psychological and health problems likely to be encountered when treating substance use disorders in Native American populations.

MICRA Project was conducted in two phases: MICRA was conducted in two phases: Phase 1 was a feasibility (N = 9) non-randomized one-group design wherein all participants received culturally adapted MICRA. The purpose of Phase 1 was to (a) implement and test the draft version of the MICRA counselor manual, (b) test counselor fidelity monitoring procedures, (c) certify counselors in MI and CRA, (d) test the assessment procedures and basic aspects of the Manual of Operations, (e) certify the research assistant in assessment administration procedures, and (e) pilot the 4- and 8-month follow-ups.

Phase 2 was a mixed efficacy/effectiveness (hybrid) randomized controlled trial of MICRA (n=38) and TAU (n=41) with a parallel design and follow-up assessments at 4-, 8-, and 12-months post baseline. Following the screening and baseline interview, participants were randomized to receive MICRA or treatment as usual (TAU). Participants randomized to MICRA could receive up to a maximum of 16 to 20 therapy sessions with one of the MICRA counselors over the course of 16 weeks. In TAU, participants received standard outpatient services at the Tribal substance use disorder treatment center.

The primary hypotheses were: (1) the feasibility test of culturally adapted MICRA (N=9) would yield improved percent days abstinent from all substances (excluding tobacco) from baseline to the 8-month follow-up, and (2) In the pilot randomized controlled trial of culturally adapted MICRA versus treatment as usual (TAU), the investigators hypothesized that percent days abstinent from all substances would be greater at the 12-month follow-up timepoint compared to TAU.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* an enrolled tribal member,
* diagnosed with a Diagnostic and Statistical Manual (DSM-IV-TR) for substance use disorder (SUD),
* seeking substance use disorder treatment
* and able to speak English fluently
* resident within the reservation or neighboring small settlements

Exclusion Criteria:

* any planned absences from reservation greater than 14 days during the 16 week treatment period,
* cannot identify at least one "locator" person for follow-up tracking,
* actively psychotic or chronic mental illness that is not well treated, or
* major cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2013-11-18 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Percent days abstinence from substances | baseline to 12-month follow-up
  using the Form-90 for drugs (Form 90-D questionnaire), the investigators will examine percent days abstinent from all substances and conduct statistical tests to determine whether there is a significant difference between the treatment and comparison conditions

SECONDARY OUTCOMES:
Condom Use Self Efficacy (questionnaire) | baseline to 12 month follow-up
  Condom Use Self-Efficacy Scale (questionnaire); the investigators will examine whether there are significant increases in condom use self-efficacy for the sample from baseline to 12-month follow-up
Native American Spirituality Scale (questionnaire) | baseline to 12 month follow-up
  The investigators will examine whether spiritual beliefs and behaviors increase over time from baseline to the 12-month follow-up for the sample using the total score as well as the two subscales (spiritual beliefs and spiritual behaviors)

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla Venner, Ph.D., Principal Investigator — University of New Mexico

IPD SHARING:
Plan to Share IPD: No
These data are owned by the tribe. If anyone would like to use these data, the PI will serve as the liaison to request permission from the tribe.

REFERENCES:
- [Background] Greenfield BL, Venner KL. Review of substance use disorder treatment research in Indian country: future directions to strive toward health equity. Am J Drug Alcohol Abuse. 2012 Sep;38(5):483-92. doi: 10.3109/00952990.2012.702170. PMID 22931083
- [Background] Venner KL, Serier K, Sarafin R, Greenfield BL, Hirchak K, Smith JE, Witkiewitz K. Culturally tailored evidence-based substance use disorder treatments are efficacious with an American Indian Southwest tribe: an open-label pilot-feasibility randomized controlled trial. Addiction. 2021 Apr;116(4):949-960. doi: 10.1111/add.15191. Epub 2020 Aug 11. PMID 32667105
- [Background] Serier KN, Venner KL, Hernandez-Vallant A. The Condom Use Self-Efficacy Scale in Substance Use Disorder Treatment-Seeking American Indian Adults. Subst Use Misuse. 2021;56(13):2066-2073. doi: 10.1080/10826084.2021.1963988. Epub 2021 Sep 30. PMID 34590538
- [Result] Greenfield BL, Hallgren KA, Venner KL, Hagler KJ, Simmons JD, Sheche JN, Homer E, Lupee D. Cultural adaptation, psychometric properties, and outcomes of the Native American Spirituality Scale. Psychol Serv. 2015 May;12(2):123-133. doi: 10.1037/ser0000019. PMID 25961648
- [Result] Venner KL, Greenfield BL, Hagler KJ, Simmons J, Lupee D, Homer E, Yamutewa Y, Smith JE. Pilot Outcome Results of Culturally Adapted Evidence-Based Substance Use Disorder Treatment with a Southwest Tribe. Addict Behav Rep. 2016 Jun 1;3:21-27. doi: 10.1016/j.abrep.2015.11.002. PMID 26951788
- [Result] Serier KN, Venner KL, Sarafin RE. Evaluating the Validity of the DSM-5 Alcohol Use Disorder Diagnostic Criteria in a Sample of Treatment-seeking Native Americans. J Addict Med. 2019 Jan/Feb;13(1):35-40. doi: 10.1097/ADM.0000000000000452. PMID 30303888

DOCUMENTS (2):
  • Study Protocol (2012-06-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT05938764/Prot_000.pdf
  • Informed Consent Form (2012-07-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT05938764/ICF_001.pdf